CLINICAL TRIAL: NCT03594422
Title: A Phase I Study to Assess the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Properties of Oral HQP1351 in Patients With GIST or Other Solid Tumors.
Brief Title: A Study of HQP1351 in Patients With GIST or Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: HealthQuest Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-0003
Record Dates: First submitted 2018-07-01; First posted 2018-07-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Stromal Tumor (GIST); Solid Tumor, Adult
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — olverembatinib

STUDY DESIGN:
Intervention Model Description: Patients will be randomized at 1:1:1 ratio into the three dose cohorts: 30 mg QOD, 40 mg QOD and 50 mg QOD.Non-randomized selected adult subjects will receive a 40 mg QOD dosing regimen. And the minor will be enrolled to the three dose cohorts: 20mg QOD, 30 mg QOD, 40 mg QOD according to the weight.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HQP1351 30mg (Experimental): 30 mg QOD(Minor subjects will be enrolled based on weight)
  Interventions: Drug: HQP1351
- HQP1351 40mg (Experimental): 40 mg QOD(Minor subjects will be enrolled based on weight)
  Interventions: Drug: HQP1351
- HQP1351 50mg (Experimental): 50 mg QOD
  Interventions: Drug: HQP1351
- HQP1351 20mg (Experimental): 20 mg QOD (Minor subjects will be enrolled based on weight)
  Interventions: Drug: HQP1351

INTERVENTIONS:
Drug: HQP1351 — HQP1351 Orally, once every other day (QOD) for consecutive 4 weeks each cycle.

SUMMARY:
This study is a Multi-center, Open-label Phase 1 Study to Determine the Recommend Phase 2 Dose (RP2D) and Evaluate PK/PD and preliminary Efficacy of HQP1351 in Patients With GIST or Other Solid Tumors.

DETAILED DESCRIPTION:
The primary objective of this phase 1 study is to determine the RP2D of HQP1351 in patients with GIST or other solid tumors. The secondary objective is to assess the safety, tolerability, PK and preliminary anti-tumor activities of HQP1351 in Patients With GIST or Other Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or not pregnant or lactating women, age≥12years.
2. Advanced and/or metastatic GIST or other solid tumors, confirmed by histology and/or cytology. GIST patients must be primary resistant to imatinib (tumor progresses within 6 months first-line imatinib treatment, or succinate dehydrogenase B (SDHB) deficient confirmed by immunohistochemistry, or NF1 mutation), OR imatinib or imatinib and at least one other TKI treatment failure (after imatinib or other TKI treatment for more than 6 months, tumor progress again after achieving tumor remission or stability).
3. ECOG≤ 2.
4. Estimated survival at least 3 months.
5. Adequate hematologic and bone marrow functions.
6. Adequate renal and liver function.
7. Heart function index:

   * Troponin(I/T) ≤ Upper Limit of Normal;
   * Ejection fraction >40%;
   * QTc interval ≤ 450 ms in male or ≤ 470 ms in female.
8. Negative serum pregnancy test (for women of childbearing potential) documented within the 24-hour prior to the first dose of investigational product.
9. Willing to use contraception by a method that is deemed effective by the investigator by Subject and their partners throughout the treatment period and for at least 30 days following the last dose of study drug.
10. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the subject prior to any study-specific procedures).
11. Willing and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Received any anti-cancer chemotherapy, biological agent treatment (e.g. Monoclonal antibody), immunotherapy (e.g. IFN) or radiotherapy with 28 days or 5 times half- time before first dose of HQP1351.
2. Received any TKIs within 14 days before first dose of HQP1351.
3. Attended any clinical trials on other drugs within 14 days before first dose of HQP1351.
4. Have not recovered (> Grade 1 by CTCAE, v. 4.0) from AEs (except alopecia) due to agents previously administered.
5. Malabsorption syndrome or other diseases that affect the absorption of oral drugs.
6. Cardiovascular diseases of clinical significance, uncontrollable or active, including but not limited to: history of myocardial infarction; unstable history of angina pectoris; a history of congestive heart failure or lower left ventricular ejection fraction (LVEF) than normal limit within 6 months; the history of atrial arrhythmias was judged by the researchers to have important clinical significance; history of ventricular arrhythmias, etc.
7. Hypertension was still poorly controlled after medication treatment (SBP > 140 mmHg and/or DBP > 90 mmHg).
8. Concurrent use any medication led to prolong QT interval.
9. Pulmonary mean arterial pressure>35 mmHg by ECHO.
10. Significant severe cardiovascular conditions during previous TKI treatment.
11. Uncontrollable hypertriglyceridemia.
12. Performed major surgery (except for intravenous catheterization or bone marrow biopsy) within 14 days of first dose of HQP1351.
13. Arterial thrombosis or embolism events such as cerebrovascular accident (including transient ischemic attack, TIA), or venous thrombosis events or pulmonary embolism within 6 months before the first dose of HQP1351 or deep vein thrombosis within 3 months before the first dose of HQP1351.
14. Brain metastasis.
15. Had other primary malignant tumors in the last three years (exception of the tumors being cured for 5 years or more, or complete removal of non-melanoma skin cancer or successful treatment of carcinoma in situ, or the controlled prostate cancer).
16. Had active, symptomatic infections (including known infections of HIV, viral hepatitis (A, B, or C)). If there is no history of infection, screening is not required.
17. Subjects who are known to be allergic to pharmaceutical ingredients or their analogs.
18. Pregnancy or lactation, or expect to be pregnant during the study period.
19. According to the judgment of the investigator or sponsor, any symptoms or disease of the subject may jeopardize the safety or safety assessment of the subject.
20. Any other condition or circumstance of that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerance | 30 days after the last dose of HQP1351
  Patients with HQP1351 treatment related adverse events (AE), serious adverse events (SAE) will be assessed according NCI CTCAE Version 4.03.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of HQP1351 on Day 1 and Day 27 post HQP1351 treatment on cycle 1. | 28 days
  Pharmacokinetic evaluation
Area under the plasma concentration versus time curve (AUC) of HQP1351 on Day 1 and Day 27 post HQP1351 treatment on cycle 1. | 28 days
  Pharmacokinetic evaluation
Anti-tumor activities of HQP1351 | 3-60 months
  Response will be evaluated every 2 cycles (8 weeks), according to the revised RECIST Guideline, Version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Professor, Principal Investigator — Sun Yat-sen University
Locations (6):
- China (6):
  - Sun-Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong general hospital, Guangzhou, Guangdong
  - Henan cancer hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College of Huazhong University of Science ang Technology, Wuhan, Hubei
  - Chinese PLA general hospital, Beijing, China, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided